CLINICAL TRIAL: NCT03208075
Title: the Regulation of Phosphorus Homeostasis by Dietary Phosphorus Intake in Normal Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Chen Jing, Professor, Huashan Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: HuashanH-2
Record Dates: First submitted 2017-07-02; First posted 2017-07-05 (Actual); Last update posted 2017-08-15 (Actual); Status verified 2017-08

CONDITIONS: Healthy
Keywords: phosphorus,diet; phosphorus; healthy subject

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Normal Phosphorus Diet (Experimental): Diet containing 1500mg of phosphorus per day
  Interventions: Other: normal diet
- Low-phosphorus Diet (Experimental): Diet containing 500mg of phosphorus per day
  Interventions: Other: low-phosphorus diet
- High-phosphorus Die (Experimental): Diet containing 2300mg of phosphorus per day
  Interventions: Other: high-phosphorus diet

INTERVENTIONS:
Other: normal diet — Diet containing 1500mg of phosphorus
  Arms: Normal Phosphorus Diet
Other: low-phosphorus diet — Diet containing 500mg of phosphorus
  Arms: Low-phosphorus Diet
Other: high-phosphorus diet — Diet containing 2300mg of phosphorus
  Arms: High-phosphorus Die

SUMMARY:
The investigators have conducted the study about the effects of normal diet and low-phosphorus diet on phosphorus homeostasis in healthy subjects, now this study is designed to explore further about the effect of high-phosphorus diet on phosphorus homeostasis.

DETAILED DESCRIPTION:
Serum phosphate concentrations are not only associated with cardiovascular and all-cause mortality in chronic kidney disease (CKD) patients, but also associated with the mortality in community population. Thus, maintaining normal serum phosphate and reducing postprandial fluctuation of serum phosphate are essential for healthy people.

The investigators have conducted a study about the effects of normal diet (phosphorus 1500mg) and low-phosphorus diet (phosphorus 500mg) on phosphorus homeostasis in healthy men. The results showed low-phosphorus diet could significantly reduce serum phosphorus and urine phosphorus level compared to normal diet. However, the levels of serum FGF23 and a-klotho were not different between these two groups.Thus, the investigators want to further explore the effects of high-phosphorus diet (phosphorus 2300mg)on phosphorus homeostasis in healthy men.

Therefore, the investigators plan to conduct a crossover clinical study to evaluate the phosphorus homeostasis modulated by native normal diet, restricted phosphorus diet, high phosphorus diet and then to explore the underlying mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 18-45 years
* Healthy volunteers: no history of chronic diseases; no active symptoms or physical signs; negative results of electrocardiogram and chest X-ray; biochemical indicators of regular medical examination are within 95%-105% of normal range.
* Willingness to sign the consent form approved by an Institutional Review Board and comply with the study protocol.
* Body mass index ranged within 18.5-24 kg/m2.

Exclusion Criteria:

* Current history of drug or alcohol abuse as assessed by the principal Investigator.
* Subject has blood donations or blood loss more than 300ml within three months
* Allergic to more than two foods or drugs.
* Subject has psycho-disability or body disability.
* Subject has a condition that in the judgment of the Principal Investigator could potentially pose a health risk to the patient while involved in the study.
* Subject has participated in the other clinical trials at the same time.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
Circadian rhythm of serum phosphorus concentration | 24 hour

SECONDARY OUTCOMES:
Circadian rhythm of urine phosphorus concentration | 24 hour
Circadian rhythm of plasma fibroblast growth factor 23 (FGF23) | 24 hour
Circadian rhythm of parathyroid hormone (PTH) | 24 hour
Circadian rhythm of 1, 25-dihydroxyvitamin D (1,25(OH)2D3) | 24 hour

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan hospital, Shanghai Medical College, Fudan University, Shanghai, Shanghai Municipality, China